CLINICAL TRIAL: NCT02313870
Title: Comparison of Monotherapy With Protracted Superpotent Topical Steroids to Superpotent Topical Steroids Associated With Methotrexate in Bullous Pemphigoid
Brief Title: Topical Steroids Alone or Associated With Methotrexate in Bullous Pemphigoid
Acronym: BP/MTX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7850
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; superpotent topical steroids; methotrexate; safety
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Clobetasol; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Superpotent topical steroids/methotrexate
  Interventions: Drug: clobetasol propionate + Methotrexate
- B (Other): Superpotent topical steroids (clobetasol propionate)
  Interventions: Drug: clobetasol propionate alone

INTERVENTIONS:
Drug: clobetasol propionate + Methotrexate — daily applications of topical clobetasol propionate at a dose of 10 to 30 g / day depending on the patient's weight and the initial number of new blisters per day, associated with methotrexate (MTX) received either orally or subcutaneously at a dose of 12.5 mg / week in patients weighing less than 60 kg and with creatinine clearance greater than 50 ml / min (planned dose reduction to 10 mg / week in patients less than 60 kg or with a creatinine clearance less than 50 ml / min) for four weeks followed by oral or subcutaneous methotrexate alone at the same dose during following 8 months
  Arms: A
Drug: clobetasol propionate alone — daily applications of topical clobetasol propionate at a dose of 10 to 30 g / day depending on the patient's weight and the initial number of new blisters per day, up to 14 days after control of the disease followed by 1 application every 2 days at the same dose for 4 weeks then an application twice a week for 4 weeks then once application a week until the end of the 9th month of treatment
  Arms: B

SUMMARY:
This controlled multi-center randomized clinical trial, with direct individual benefit, will compare efficacy and safety of two strategies in non-localized BP care: a combined regimen using initial superpotent topical steroids associated with methotrexate for 4 weeks followed by methotrexate alone for 8 months and superpotent topical steroids alone maintained 9 months (current standard of care). The expected result is an equivalence between the two compared strategies in terms of safety and efficacy, MTX monotherapy during the maintenance phase being easier to manage and therefore associated with better compliance than topical steroids with less cutaneous side effects and most cost-effective.

DETAILED DESCRIPTION:
Bullous pemphigoid (BP) is a rare mucocutaneous autoimmune bullous disorder (incidence <1/10000 / year in France) that mostly affects elderly patients. Its mortality rate is as high as 20 to 40% at one year. A study initiated by the French group for bulllous disorders devoted to the study of autoimmune bullous diseases the study of autoimmune bullous diseases and which is an international leader on this issue, has previously demonstrated the efficacy and relatively good tolerance of superpotent topical corticosteroids in BP.However, the use of superpotent topical corticosteroids is flawed with practical difficulties (home-based care by nurses once or twice a day to administer treatment, this for several months) and its cost is significantly higher than that an oral steroid treatment as a consequence. On the other hand, there is probably a non-negligible systemic absorption of superpotent topicalsteroid responsible for potentially serious side effects similar to those encountered with systemic corticosteroids. Finally, a protracted treatment with superpotent topical steroid most often causes skin atrophy with deleterious consequences.It would then be of interest to be able to significantly reduce the duration of use of topical steroids through an early-associated systemic treatment relying on an easy-to-use and relatively safe molecule that would maintain the disease under control after an initial clinical remission has been achieved by initial and time-limited use of superpotent topical steroids. Methotrexate (MTX) could be an interesting candidate in this regard, with a low-level and tolerable short- and middle-term toxicity if small doses are used (10-15 mg / week) while its long-term safety is usually irrelevant in elderly patients. Its use and monitoring are relatively easy and a number of international publications, including two recent French ones, have shown efficacy in this setting including a relaying strategy after initial use of superpotent topical steroids in BP treatment, in preliminary open studies .These encouraging results prompt to propose a controlled multi-center randomized clinical trial, with direct individual benefit, comparing efficacy and safety of a treatment regimen using superpotent topical steroids alone maintained 9 months (current standard of care) to a mixed initial treatment combining applications of superpotent topical steroids associated with methotrexate for 4 weeks followed by methotrexate alone for 8 additional months in non-localized BP. In both arms, the total treatment duration will then be 9 months. The two arms of the study will be:Arm A: daily applications of topical clobetasol propionate at a dose of 10 to 30 g / day depending on the patient's weight and the initial number of new blisters per day, associated with methotrexate (MTX) received either orally or subcutaneously at a dose of 12.5 mg / week in patients weighing less than 60 kg and with creatinine clearance greater than 50 ml / min (planned dose reduction to 10 mg / week in patients less than 60 kg or with a creatinine clearance less than 50 ml / min) for four weeks followed by oral or subcutaneous methotrexate alone at the same dose during following 8 monthsArm B: daily applications of topical clobetasol propionate at a dose of 10 to 30 g / day depending on the patient's weight and the initial number of new blisters per day maintained until 14 days after full disease control followed by the same daily dose applied every other day for a month and then twice a week for a month and then once a week until the end of the 9th month.The primary endpoint will be the actuarial survival rate at one year in both groups and secondary endpoints will be the initial control rate of the disease, the number of serious side effects during treatment and the number of relapses during treatment.The expected result is an equivalence between the two compared strategies in terms of safety and efficacy, MTX monotherapy during the maintenance phase being easier to manage and therefore associated with better compliance than topical steroids with less cutaneous side effects and most cost-effective.This study will enroll 150 patients per arm and will include a follow up of 9 months with 9 visits per patient.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years old or more
* Patients affiliated to social security system,
* Bullous pemphigoid diagnosed according to the following criteria: presence of at least 3 of the 4 clinical criteria for bullous pemphigoid as published by the french group for study of blistering diseases (positive predictive value: 95 %: age over 70 years, no lesions on neck or head, absence of atrophic scars, no mucosal lesions.= Histological Examination consistent with BP diagnosis and carried out in the month before inclusion: existence of a sub epidermal blister regardless of its size, containing neutrophils and / or eosinophils associated with a dermal infiltrate consisting of neutrophils and / or eosinophils, or to margination of neutrophils and / or eosinophils along the dermoepidermal junction.= Direct immunofluorescence performed (DIF) in the month preceding inclusion and showing linear deposition of IgG and / or C3 along the dermo-epidermal junction.
* Patients: = no prior topical steroid or superpotent topical steroids for less than 16 days using the same or equivalent dosage as the one used in the study a different regimen and this regardless of the clinical resultsOR receiving potent or superpotent topical steroids for at least 16 days with a different regimen than that used during the trial AND not controlled by this treatment (appearance of at least 3 new blisters per day)
* written consent of the patient or, if not possible, certified by a third party,
* effective contraception (oral or intrauterine device) set up at least one month before inclusion for women of childbearing age,
* For women of reproductive age (age <50 years), negative serum pregnancy test at inclusion
* Serum albumin ≥ 25 g / L

Exclusion Criteria:

* Localized bullous pemphigoid (area <400 cm2: 20 x 20 cm)
* Major blood cytopenia: Hb ≤ 10 g / dl and / or leukocytes ≤ 3000 / mm3 and / or platelets ≤ 100,000 / mm3
* Creatinine Clearance appreciated by the formula MDRD <30 ml / min
* Serum albumin <25 g / L
* pregnancy-associated Pemphigoid
* Linear IgA Dermatosis identified by DIF
* Pemphigoid with clinically dominant mucosal lesions
* Relapse of previously diagnosed pemphigoid and still receiving treatment or for whom treatment was stopped for less than six months
* Known allergy to topical steroids and / or methotrexate
* recent history of liver disease (within two years) regardless of its nature or presence of active liver disease (transaminases and / or alkaline phosphatase greater than twice the upper standard laboratory)
* Chronic alcoholism (declared consumption of more than 60 g alcohol / day or approximately 0.5 L / day of wine)
* patient receiving notoriously hepatotoxic drugs or that can interfere with metabolism or haematological toxicity of Methotrexate
* Peptic ulcer proven by endoscopy performed during the last 15 days
* Severe Active infection regardless of its nature
* Evolutive neoplasia whatever its nature except basal cell carcinoma
* Poorly controlled diabetes mellitus (fasting glucose greater than or equal to 2 2.5 g / L and / or Hb A1C greater than or equal to 8.5% before treatment)
* disease that can not be possibly monitored on a regular basis
* acquired or congénital Immunosuppression
* known HIV Seropositivity
* Chronic respiratory failure
* Pregnancy or breastfeeding
* Patient of childbearing age and not using effective contraception
* Patient incapable of giving informed consent and for whom a family member or a trustworthy third party does not grant participation in the study, protected adults, vulnerable people (art. L1121-6, L1121-7, L 1121-8, L1121-9) or patient accrued in another clinical research study
* Long-term treatment prescribed for another illness by steroids, immunosuppressive drugs, cyclosporin or any other treatment that may have been successfully used in the treatment of bullous pemphigoid (dapsone, Gamma globulins, plasma exchange, tetracyclines). For all previous medications, a minimum clearance of two months is required before enrollment in the present trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-01-22 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
actuarial survival | 9 months
  The primary endpoint is the actuarial survival rate with or without recurrence at 9 months in the topical steroid + methotrexate group (Arm A) compared to exclusive topical steroid group (Arm B).

SECONDARY OUTCOMES:
Initial control rate of the disease | 9 months
  The initial control rate of the disease at D28 (Visit 4)
Safety: The frequency of serious and significant adverse events | 9 months
Frequency of relapses | 9 months
  The frequency of relapses during treatment
Relapse-free survival | 9 months
  relapse-free survival
Easiness of use | 9 months
  Easiness of use indirectly estimated by treatment complicance evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Dereure, MD, PhD, Principal Investigator — University of Montpellier France; French Society of Dermatology; french group for study of blistering diseases
Locations (1):
- University Hospital Of Montpellier, Montpellier, France